CLINICAL TRIAL: NCT02147067
Title: Microvascular Assessment of Ranolazine in Non-Obstructive Atherosclerosis
Brief Title: Microvascular Assessment of Ranolazine in Non-Obstructive Atherosclerosis (MARINA)
Acronym: MARINA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Habib Samady, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00072996
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Microvascular Angina
Keywords: microvascular angina; coronary microvascular disease; coronary physiology; ranolazine
MeSH Terms: conditions — Microvascular Angina | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ranolazine (Experimental): Ranolazine 1,000 mg twice daily
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 1,000 mg twice daily
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at the effects of the drug Ranolazine compared to Placebo on symptoms of chest pain or chest tightness (known as angina), exercise endurance and ability, and changes in blood flow to the very small arteries of the heart (known as coronary microvascular function) in patients who do not have significant blockages in their major heart arteries. Ranolazine is a drug that is already approved by the FDA for angina, but it may be particularly effective in people with disease in their tiny heart vessels (known as coronary microvascular disease).

This trial aims to enroll 50 patients with angina who undergo baseline bicycle exercise testing with monitoring of the heart's electrical activity and oxygen consumption (known as cardiopulmonary exercise test) and coronary angiogram (taking pictures of the heart arteries through small hollow tubes placed through the wrist or groin). If severe blockages in the main arteries are not found then testing for coronary microvascular function will be performed. Subsequently, participants will then be randomized 50/50 to either Ranolazine or Placebo. After taking the study drug for 12 weeks, they will then repeat the cardiopulmonary exercise test and the coronary angiogram with testing for microvascular function.

DETAILED DESCRIPTION:
Heart disease is the most common cause of death in the world. Most of our understanding of heart disease has involved the large heart arteries (epicardial arteries); however, disease of the very small heart arteries (coronary microvasculature) likely precedes the development of epicardial disease and represents the "base of the iceberg" of cardiovascular disease. Yet, we do not understand how dysfunctional microvasculature leads to reduced blood flow, symptoms and adverse outcomes.

Coronary microvascular disease results from a combination of structural and functional abnormalities, so it is important to have reliable diagnostic tools that do not rely solely on imaging. The gold-standard for testing involves hemodynamic (blood circulation) measurements such as coronary flow reserve (CFR) and hyperemic microcirculatory resistance (HMR) that take place in the cardiac catheterization laboratory.

Ranolazine is a relatively new U.S Food and Drug Administration-approved medicine to help with angina (chest pain). There are no publications on the effect of Ranolazine on HMR.

ELIGIBILITY:
Inclusion Criteria:

* History of typical angina or effort-induced anginal symptoms and are currently experiencing angina at least once per week
* Abnormal stress ECG, exercise stress imaging, or pharmacological stress imaging
* Non-obstructive coronary artery disease as defined by lesion stenosis ≤ 50% in any artery as visualized by diagnostic angiography

Exclusion Criteria:

* Inability to provide informed consent
* Active Myocardial Infarction
* History of coronary artery bypass grafting
* Diagnosis of other specific cardiac disease such as severe valvular heart disease, cardiomyopathy, or variant angina
* Left Ventricular Ejection Fraction (LVEF) < 30%
* Known renal insufficiency (CrCl < 30 mL/min) or on dialysis
* Contraindications to the use of Ranolazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Samady, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Koh JS, Hung OY, Eshtehardi P, Kumar A, Rabah R, Raad M, Kumar S, Chaudhry S, Gupta S, Hosseini H, Brilakis E, Corban M, Sabbak N, Burnett GM, Liu C, Mehta PK, Quyyumi AA, Samady H. Microvascular Assessment of Ranolazine in Non-Obstructive Atherosclerosis: The MARINA Randomized, Double-Blinded, Controlled Pilot Trial. Circ Cardiovasc Interv. 2020 Dec;13(12):e008204. doi: 10.1161/CIRCINTERVENTIONS.119.008204. Epub 2020 Dec 4. PMID 33272036
- [Derived] Titterington JS, Hung OY, Wenger NK. Microvascular angina: an update on diagnosis and treatment. Future Cardiol. 2015 Mar;11(2):229-42. doi: 10.2217/fca.14.79. PMID 25760881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital in Atlanta, Georgia. Participant enrollment began in September 2014 and all study procedures were completed in June 2018.
Groups:
- Ranolazine: Participants receiving 500mg twice a day for 2 weeks then 1000mg twice daily of ranolazine for 10 weeks
- Placebo: Participants receiving a placebo to match the ranolazine dose for 12 weeks
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 13 | 13
Completed | 11 | 11
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants completing the study are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.3) | 51.9 (13.9) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 7 | 15
  African American | 2 | 3 | 5
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22
Hypertension [Count of Participants; unit: Participants] | 8 | 8 | 16
Prior myocardial infarction [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Seattle Angina Questionnaire Score Regarding Angina Frequency
Description: The change in scores of the angina frequency dimension of the Seattle Angina Questionnaire (SAQ) after 12 weeks therapy with ranolazine or placebo are presented. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Individual dimensions of the Seattle Angina Questionnaire are transformed to be a score from 0 to 100, where higher scores indicate better health. A positive number for the angina frequency dimension means that the participants are experiencing fewer episodes of angina at week 12 than they were at the baseline visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 0.70 (1.26) | 0.27 (0.62)

2. Secondary Outcome: Change in Seattle Angina Questionnaire Score Regarding Physical Limitation
Description: The change in scores of the physical limitation dimension of the Seattle Angina Questionnaire (SAQ) after 12 weeks therapy with ranolazine or placebo are presented. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Individual dimensions of the Seattle Angina Questionnaire are transformed to be a score from 0 to 100, where higher scores indicate better health. A positive number for the physical limitation dimension means that the participants are experiencing less limitation at week 12 than they were at the baseline visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | -0.09 (0.25) | 0.27 (0.68)

3. Secondary Outcome: Change in Seattle Angina Questionnaire Score Regarding Angina Stability
Description: The change in scores of the angina stability dimension of the Seattle Angina Questionnaire (SAQ) after 12 weeks therapy with ranolazine or placebo are presented. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Individual dimensions of the Seattle Angina Questionnaire are transformed to be a score from 0 to 100, where higher scores indicate better health. A positive number for the angina stability dimension means that the participants are experiencing fewer changes in their angina at week 12 than they were at the baseline visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 0.00 (0.79) | 0.50 (1.16)

4. Secondary Outcome: Change in Seattle Angina Questionnaire Score Regarding Treatment Satisfaction
Description: The change in scores of the treatment satisfaction dimension of the Seattle Angina Questionnaire (SAQ) after 12 weeks therapy with ranolazine or placebo are presented. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Individual dimensions of the Seattle Angina Questionnaire are transformed to be a score from 0 to 100, where higher scores indicate better health. A positive number for the treatment satisfaction dimension means that the participants are experiencing greater satisfaction with their treatment at week 12 than they were at the baseline visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 1.17 (3.92) | 0.28 (0.49)

5. Secondary Outcome: Change in Seattle Angina Questionnaire Score Regarding Disease Perception
Description: The change in scores of the disease perception dimension of the Seattle Angina Questionnaire (SAQ) after 12 weeks therapy with ranolazine or placebo are presented. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Individual dimensions of the Seattle Angina Questionnaire are transformed to be a score from 0 to 100, where higher scores indicate better health. A positive number for the disease perception dimension means that the participants felt that their disease impacted their quality of life less at week 12 than at the baseline visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 0.89 (1.49) | 1.00 (0.99)

6. Secondary Outcome: Change in Peak Rate of Oxygen Consumption (VO2 Max)
Description: The change in VO2, as measured by cardiopulmonary exercise testing (CPET), after 12 weeks therapy with ranolazine compared with placebo. VO2 max is the maximum amount of oxygen the participants are utilizing during intense treatment. To standardize exercise stress testing, CPET was performed under the guidance of the MET-TEST CPET network in Atlanta, Georgia. The MET-TEST was created in 2003 and is a high-precision stress test with detailed physiological assessment, allowing accurate and reproducible measurements of peak VO2. Individuals may demonstrate an abnormal CPET response before they develop symptoms or present with cardiac events and abnormal CPET results are strong predictors of future adverse outcomes. Higher VO2 values indicate better oxygen utility and positive value for VO2 change means there was improvement from baseline at the week 12 visit. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
L/min | -0.03 (0.23) | 0.06 (0.11)

7. Secondary Outcome: Change in Time to Angina
Description: Change in time to angina as measured by cardiopulmonary exercise testing after 12 weeks therapy with Ranolazine compared with placebo. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline.
Time Frame: Baseline, Week 12
Population: Data for this outcome measure was not collected.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Metabolic Equivalents of Task (METs) at Peak
Description: Change in exercise was measured as Metabolic Equivalents of Task (METs) at Peak by cardiopulmonary exercise testing (CPET) after 12 weeks therapy with ranolazine compared with placebo. METs are used to describe functional aerobic capacity and harder physical tasks require a higher number of METs. METs at a peak level of exercise was determined for each participant. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. A positive value for change in METs at Peak of exercise indicates that the participant has improved their aerobic capacity from baseline at the week 12 visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: 3.5ml of oxygen/kg per min
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
3.5ml of oxygen/kg per min | 0.00 (0.20) | 4.42 (14.45)

9. Secondary Outcome: Change in Coronary Flow Reserve (CFR)
Description: The changes in Coronary Flow Reserve (CFR) after 12 weeks therapy with ranolazine compared with placebo are presented here. CFR is a measurement of the maximum increase of blood flow through the coronary arteries during exercise. Average peak velocity (APV) was assessed over a 3- to 5-beats period. CFR was defined as the ratio of hyperemic to basal APV. A low CFR is an indication of coronary artery disease. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. A positive value for the change in CFR suggests improvement in coronary artery blood flow between the baseline and week 12 visits.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: ratio of hyperemic to basal APV
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
ratio of hyperemic to basal APV | 0.38 (0.85) | 0.09 (0.30)

10. Secondary Outcome: Change in Hyperemic Microcirculatory Resistance (HMR)
Description: Change in Hyperemic Microcirculatory Resistance (HMR) after 12 weeks therapy with ranolazine compared with placebo. Average peak velocity (APV) was assessed over a 3- to 5-beats period. HMR was measured as the ratio of distal pressure to APV. Change at 12 weeks was calculated as (Endpoint Value at 12 weeks - Endpoint Value at Baseline)/Endpoint Value at Baseline. Higher HMR is associated with myocardial ischemia and a positive value for change in HMR indicates increased risk for cardiac events at the week 12 visit.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mmHg/cm/s
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 11 | 11
mmHg/cm/s | 0.14 (0.50) | -0.04 (0.42)

11. Secondary Outcome: Percent Change in Coronary Blood Flow
Description: Coronary endothelial function will also be evaluated by measurement of coronary blood flow during infusion of intracoronary acetylcholine. Coronary blood flow (CBF) is defined as diameter (D)2 x APV / 8. Percent change in CBF (%ΔCBF) is calculated by (CBFACh - CBFbaseline) / CBFbaseline x 100%, where a >50% increase in CBF in response to acetylcholine is considered normal.
Time Frame: Baseline, Week 12
Population: Data for this outcome measure was not collected.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study enrollment until completion of follow-up (12 weeks)
Description: The study investigators will record adverse effects, whether anticipated or unanticipated. All adverse events will be captured on an adverse event case report form and tracked from time of study enrollment until completion of all study follow-up (12 weeks).
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT02147067/Prot_SAP_000.pdf